CLINICAL TRIAL: NCT04392323
Title: Incidence of COVID-19 Test Conversion in Post-surgical Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Northwell Health (Other)
Responsible Party: Principal Investigator, Ernesto Molmenti, Vice Chairman of Surgery - Chief of Innovation. North Shore University Hospital, Northwell Health. Professor of Surgery, Medicine, and Pediatrics, Zucker School of Medicine at Hofstra/Northwell, Northwell Health
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: IRB #20-0404
Record Dates: First submitted 2020-05-15; First posted 2020-05-18 (Actual); Last update posted 2021-11-08 (Actual); Status verified 2020-05

CONDITIONS: Sars-CoV2
Keywords: Sars-CoV2; surgery; infection; transmission; Covid-19; safety; nosocomial; virus; corona; COVID; incidence
MeSH Terms: conditions — Infections; COVID-19; Virus Diseases

STUDY DESIGN:
Intervention Model Description: Prospective Cohort
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Study Group (Experimental): Patients will be recruited as an outpatient prior to their surgical procedure or during their hospital admission. If they consent, they will provide signed informed consent and will receive testing with serology and PCR for COVID-19 infection at pre-surgical testing 24-48 hours prior to their scheduled procedure. If they consent while inpatient postoperatively, signed informed consent will be procured after they have completed their pre-operative COVID-19 testing. PCR for COVID entails obtaining a nasopharyngeal swab to determine whether there is active viral replication and viral shedding. They will then have a second test with serology and PCR for COVID-19 infection 12-16 days after discharge from the hospital.
  Interventions: Diagnostic Test: COVID-19 PCR and Serology

INTERVENTIONS:
Diagnostic Test: COVID-19 PCR and Serology — PCR for COVID entails obtaining a nasopharyngeal swab (a cotton tip introduced via the nose to obtain a sample) to determine whether there is active viral replication and viral shedding. They will then have a second test with serology and PCR for COVID-19 infection 12-16 days after discharge from the hospital. Serology implies that a blood sample will be obtained by venipuncture. A volume of 50 ml (about 4 tablespoons) or less of blood will be obtained.

SUMMARY:
The current Sars-CoV-2 (COVID-19) pandemic has created major changes in how physicians perform routine healthcare for our patients, including elective and non-elective surgical procedures. Beginning on March 16th, 2020 Northwell Health postponed all elective surgeries. As the incidence of COVID-19 cases begins to decrease and hospital volume improves we need to ensure the safety of our patients planning surgical procedures. However, at this time there is a scarcity of data regarding the COVID-19 test conversion rate in surgical patients. Our goal is to determine the COVID-19 test conversion rate in these patients to better guide strategies for restarting surgical care in a large-scale pandemic.

Patients will be routinely tested with serology and PCR for COVID-19 24-48 hours prior to their scheduled surgery. Those who provide informed consent will be re-tested 12-16 days after discharge from the hospital to determine any potential nosocomial infection rate. Patients will also answer a few questions during their retest to allow the study team to gauge exposure risk postoperatively after leaving the hospital.

DETAILED DESCRIPTION:
The rapid spread of the COVID-19 infection has led to a near global lockdown including a pause in all elective surgeries [1-6]. Multiple healthcare systems and surgical societies recommended ceasing all elective procedures until this crisis is contained [7-10]. As such, it will be necessary for hospitals to restructure as surgeries increase to protect surgical patients from becoming infected. Our study will be the first to define the test conversion rate of those undergoing surgical procedures during the COVID-19 pandemic. The information gathered from this study can have implications in how surgical centers treat patients during and after this pandemic.

There has been a single study examining postoperative nosocomial infections during the initial incubation period in which 100% of patients developed Sars-CoV-2 viral pneumonia, 14 (44%) required ICU admission with mechanical ventilation, and 7 (20.5%) died after ICU admission [11]. A second cohort of bariatric surgery patients found that 4 of 4 (100%) developed Sars-CoV-2 infections postoperatively with all patients surviving [12]. Another retrospective study found that of 305 patients admitted to the digestive surgery service, 15 (4.9%) developed nosocomial Sars-CoV-2 pneumonia [13]. Of this cohort, two patients died, and seven were hospitalized with six discharged at the time of chart review. Another retrospective non-operative hospital cohort found that 34 of 102 adult patients contracted Sars-CoV-2 as a nosocomial infection. In a review of Gynecologic Oncology procedures in Wuhan the overall nosocomial infection rate was 1.59% (3/189) with two of the three patients being discharged by the publication date [14]. However, in a retrospective review of a general hospital ward in Hong Kong in which the staff used 'vigilant basic infection control measures' 10 patients and 7 staff members that met the definition for close contact were identified and through contact tracing 76 tests were performed on 52 contacts with no Sars-CoV-2 infections identified [15]. Another cohort from Wuhan demonstrated that when performing regional anesthesia (45/49 for Cesarean Section), no anesthetists were infected when complying with level 3 PPE [16].

1. Huang C, Wang Y, Li X, et al. Clinical features of patients infected with 2019 novel coronavirus in Wuhan, China. Lancet 2020;395:497-506.
2. Guan, Wei-jie, et al. "Clinical characteristics of coronavirus disease 2019 in China." New England journal of medicine (2020).
3. Wu JT, Leung K, Leung GM. Nowcasting and forecasting the potential domestic and international spread of the 2019-nCoV outbreak originating in Wuhan, China: a modelling study. Lancet 2020 January 31 (Epub ahead of print).
4. Li Q, Guan X, Wu P, et al. Early transmission dynamics in Wuhan, China, of novel coronavirus-infected pneumonia. N Engl J Med. DOI: 10.1056/NEJMoa2001316.
5. Hanna, T.P., Evans, G.A. and Booth, C.M., 2020. Cancer, COVID-19 and the precautionary principle: prioritizing treatment during a global pandemic. Nature Reviews Clinical Oncology, 17(5), pp.268-270.
6. Brindle, M. and Gawande, A., 2020. Managing COVID-19 in surgical systems. Annals of Surgery.
7. American College of Surgeons (2020). COVID-19: Recommendations for Management of Elective Surgical Procedures. Retrieved March 13, 2020 from https://www.facs.org/covid-19/clinical-guidance/elective-surgery
8. SAGES (2020). SAGES AND EAES RECOMMENDATIONS REGARDING SURGICAL RESPONSE TO COVID-19 CRISIS. Retrieved March 29, 2020 from https://www.sages.org/recommendations-surgical-response-covid-19/
9. American Society of Plastic Surgeons (2020). APS Guidance Regarding Elective and Non-Essential Patient Care. Retrieved March 19th , 2020 from https://www.plasticsurgery.org/for-medical-professionals/covid19-member-resources/previous-statements
10. American College of Obstetrics and Gynecology (2020). Joint Statement: Scheduling Elective Surgeries. Retrieved March 16th, 2020 from https://www.sgo.org/clinical-practice/management/scheduling-elective-surgeries/
11. S. Lei, F. Jiang, W. Su, et al.Clinical characteristics and outcomes of patients undergoing surgeries during the incubation period of COVID-19 infection. EClinicalMedicine (2020), p. 100331
12. Aminian A, Kermansaravi M, Azizi S, et al. Bariatric Surgical Practice During the Initial Phase of COVID-19 Outbreak [published online ahead of print, 2020 Apr 20]. Obes Surg. 2020;1-4. doi:10.1007/s11695-020-04617-x
13. Luong-Nguyen M, Hermand H, Abdalla S, et al. Nosocomial infection with SARS-CoV-2 within Deparments of Digestive Surgery. [published ahead of print, 2020 Apr 27] J of Vis Surg. 2020.
14. Yang S, Zhang Y, Cai J, Wang Z. Clinical Characteristics of COVID-19 After Gynecologic Oncology Surgery in Three Women: A Retrospective Review of Medical Records [published online ahead of print, 2020 Apr 7]. Oncologist. 2020;10.1634/theoncologist.2020-0157. doi:10.1634/theoncologist.2020-0157
15. Wong SC, Kwong RT, Wu TC, et al. Risk of nosocomial transmission of coronavirus disease 2019: an experience in a general ward setting in Hong Kong [published online ahead of print, 2020 Apr 4]. J Hosp Infect. 2020; doi:10.1016/j.jhin.2020.03.036
16. Zhong Q, Liu YY, Luo Q, et al. Spinal anaesthesia for patients with coronavirus disease 2019 and possible transmission rates in anaesthetists: retrospective, single-centre, observational cohort study [published online ahead of print, 2020 Mar 28]. Br J Anaesth. 2020;S0007-0912(20)30161-6. doi:10.1016/j.bja.2020.03.007

ELIGIBILITY:
Inclusion Criteria:

1. Patients of any ethnic background undergoing an elective surgical procedure with a minimum of 24-hour hospital admission.
2. Age ≥18.
3. Written Voluntary Informed Consent.

Exclusion Criteria:

1. Patients age < 18 years.
2. Prior documented COVID-19 Infection.
3. Current hospital inpatient prior to procedure.
4. Person Under Investigation for COVID-19 infection.
5. Current use of antiviral medications.
6. Severe or uncontrolled, concurrent medical disease (e.g. uncontrolled diabetes, unstable angina, myocardial infarction within 6 months, congestive heart failure, etc.) .
7. Documented immunodeficiency.
8. Patients with dementia or altered mental status that would prohibit the giving and understanding of informed consent at the time of study entry.
9. Outpatient procedures with planned same-day discharge.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 111 (Actual)
Dates: Start 2020-05-13 (Actual); Primary Completion 2020-10-01 (Actual); Study Completion 2020-10-04 (Actual)

PRIMARY OUTCOMES:
COVID-19 Test Conversion | 14 days
  Patients that have negative pre-operative testing that convert to positive testing 14 days post-discharge

SECONDARY OUTCOMES:
Duration of Hospitalization | 14 days
  Days from hospital admission to discharge.
Rate of self-reported COVID-19 exposure | 14 days
  Patients will be asked to describe if they have had any exposure to COVID-19 positive persons after their hospital stay.
Rate of complications from COVID-19 | 14 days
  If patients contract COVID-19 during the postoperative period, what complications occur?

CONTACTS AND LOCATIONS:
Overall Officials: Ernesto Molmenti, MD, PhD, MBA, Principal Investigator — Northwell Health; Aaron Nizam, MD, Principal Investigator — Northwell Health
Locations (2):
- United States (2):
  - North Shore University Hospital, Manhasset, New York
  - Long Island Jewish Medical Center, New Hyde Park, New York

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Huang C, Wang Y, Li X, Ren L, Zhao J, Hu Y, Zhang L, Fan G, Xu J, Gu X, Cheng Z, Yu T, Xia J, Wei Y, Wu W, Xie X, Yin W, Li H, Liu M, Xiao Y, Gao H, Guo L, Xie J, Wang G, Jiang R, Gao Z, Jin Q, Wang J, Cao B. Clinical features of patients infected with 2019 novel coronavirus in Wuhan, China. Lancet. 2020 Feb 15;395(10223):497-506. doi: 10.1016/S0140-6736(20)30183-5. Epub 2020 Jan 24. PMID 31986264
- [Result] Guan WJ, Ni ZY, Hu Y, Liang WH, Ou CQ, He JX, Liu L, Shan H, Lei CL, Hui DSC, Du B, Li LJ, Zeng G, Yuen KY, Chen RC, Tang CL, Wang T, Chen PY, Xiang J, Li SY, Wang JL, Liang ZJ, Peng YX, Wei L, Liu Y, Hu YH, Peng P, Wang JM, Liu JY, Chen Z, Li G, Zheng ZJ, Qiu SQ, Luo J, Ye CJ, Zhu SY, Zhong NS; China Medical Treatment Expert Group for Covid-19. Clinical Characteristics of Coronavirus Disease 2019 in China. N Engl J Med. 2020 Apr 30;382(18):1708-1720. doi: 10.1056/NEJMoa2002032. Epub 2020 Feb 28. PMID 32109013
- [Result] Wu JT, Leung K, Leung GM. Nowcasting and forecasting the potential domestic and international spread of the 2019-nCoV outbreak originating in Wuhan, China: a modelling study. Lancet. 2020 Feb 29;395(10225):689-697. doi: 10.1016/S0140-6736(20)30260-9. Epub 2020 Jan 31. PMID 32014114
- [Result] Li Q, Guan X, Wu P, Wang X, Zhou L, Tong Y, Ren R, Leung KSM, Lau EHY, Wong JY, Xing X, Xiang N, Wu Y, Li C, Chen Q, Li D, Liu T, Zhao J, Liu M, Tu W, Chen C, Jin L, Yang R, Wang Q, Zhou S, Wang R, Liu H, Luo Y, Liu Y, Shao G, Li H, Tao Z, Yang Y, Deng Z, Liu B, Ma Z, Zhang Y, Shi G, Lam TTY, Wu JT, Gao GF, Cowling BJ, Yang B, Leung GM, Feng Z. Early Transmission Dynamics in Wuhan, China, of Novel Coronavirus-Infected Pneumonia. N Engl J Med. 2020 Mar 26;382(13):1199-1207. doi: 10.1056/NEJMoa2001316. Epub 2020 Jan 29. PMID 31995857
- [Result] Hanna TP, Evans GA, Booth CM. Cancer, COVID-19 and the precautionary principle: prioritizing treatment during a global pandemic. Nat Rev Clin Oncol. 2020 May;17(5):268-270. doi: 10.1038/s41571-020-0362-6. PMID 32242095
- [Result] Brindle ME, Gawande A. Managing COVID-19 in Surgical Systems. Ann Surg. 2020 Jul;272(1):e1-e2. doi: 10.1097/SLA.0000000000003923. No abstract available. PMID 32209891
- [Result] Lei S, Jiang F, Su W, Chen C, Chen J, Mei W, Zhan LY, Jia Y, Zhang L, Liu D, Xia ZY, Xia Z. Clinical characteristics and outcomes of patients undergoing surgeries during the incubation period of COVID-19 infection. EClinicalMedicine. 2020 Apr 5;21:100331. doi: 10.1016/j.eclinm.2020.100331. eCollection 2020 Apr. PMID 32292899
- [Result] Aminian A, Kermansaravi M, Azizi S, Alibeigi P, Safamanesh S, Mousavimaleki A, Rezaei MT, Faridi M, Mokhber S, Pazouki A, Safari S. Bariatric Surgical Practice During the Initial Phase of COVID-19 Outbreak. Obes Surg. 2020 Sep;30(9):3624-3627. doi: 10.1007/s11695-020-04617-x. PMID 32314249
- [Result] Luong-Nguyen M, Hermand H, Abdalla S, Cabrit N, Hobeika C, Brouquet A, Goere D, Sauvanet A. Nosocomial infection with SARS-Cov-2 within Departments of Digestive Surgery. J Visc Surg. 2020 Jun;157(3S1):S13-S18. doi: 10.1016/j.jviscsurg.2020.04.016. Epub 2020 Apr 27. PMID 32381426
- [Result] Yang S, Zhang Y, Cai J, Wang Z. Clinical Characteristics of COVID-19 After Gynecologic Oncology Surgery in Three Women: A Retrospective Review of Medical Records. Oncologist. 2020 Jun;25(6):e982-e985. doi: 10.1634/theoncologist.2020-0157. Epub 2020 Apr 7. PMID 32259322
- [Result] Wong SCY, Kwong RT, Wu TC, Chan JWM, Chu MY, Lee SY, Wong HY, Lung DC. Risk of nosocomial transmission of coronavirus disease 2019: an experience in a general ward setting in Hong Kong. J Hosp Infect. 2020 Jun;105(2):119-127. doi: 10.1016/j.jhin.2020.03.036. Epub 2020 Apr 4. PMID 32259546
- [Result] Zhong Q, Liu YY, Luo Q, Zou YF, Jiang HX, Li H, Zhang JJ, Li Z, Yang X, Ma M, Tang LJ, Chen YY, Zheng F, Ke JJ, Zhang ZZ. Spinal anaesthesia for patients with coronavirus disease 2019 and possible transmission rates in anaesthetists: retrospective, single-centre, observational cohort study. Br J Anaesth. 2020 Jun;124(6):670-675. doi: 10.1016/j.bja.2020.03.007. Epub 2020 Mar 28. PMID 32234250
- [Derived] Nizam A, Nimaroff ML, Menzin AW, Goldberg GL, Miyara SJ, Molmenti E. Nosocomial COVID-19 infection in women undergoing elective cesarean delivery: a prospective cohort study. Am J Obstet Gynecol MFM. 2022 Jan;4(1):100490. doi: 10.1016/j.ajogmf.2021.100490. Epub 2021 Sep 17. PMID 34543753